CLINICAL TRIAL: NCT06915090
Title: FIT-COACH: Fitbit Intervention With Coordinated Health Coaching and PCP Support
Acronym: FIT-COACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Jamie Faro, Assistant Professor, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00002177
Record Dates: First submitted 2025-03-25; First posted 2025-04-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: GLP - 1; Diabetes; Obesity and Obesity-related Medical Conditions; Cardiovascular Diseases
Keywords: GLP-1; Diabetes; Obesity; Health Coach; Physical Activity; Body Composition
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLP-1/Coaching Arm (Experimental): Patients enrolled in this arm will complete assessments at baseline and 3-months, and receive a 12-week health coaching intervention (up to 6 virtual sessions with health coach) in addition to a Fitbit wearable device.
  Interventions: Behavioral: Health Coach/Fitbit

INTERVENTIONS:
Behavioral: Health Coach/Fitbit — Health coach visits (up to 6) will be conducted virtually and include:
  Session 1:
  * Assessment, wellness vision,
  * Habits and goals (Stretching, strength training, cardiovascular PA/walking, Diet)
  * Motivation, resources, and guidelines
  * Online program orientation
  * Set first week's goals
  Sessions 2-5:
  -Goal review, successes and challenges, new goal setting (i.e. Increase steps by 1,000/day if consistently meeting goal)
  Session 6
  -Review of progress, maintenance plan, final assessment

SUMMARY:
In individuals with overweight/obesity, increases in physical activity (PA) can improve metabolic and cardiovascular health, independent of weight loss. However, PA levels are often low in individuals with overweight/obesity, and primary care providers (PCPs) are tasked with addressing this issue. The investigative team developed and successfully piloted integrating a Fitbit program into clinical care, where patients were referred by PCPs, and PCPs could view PA data in the Epic electronic health record. Though feasible, PCPs wanted additional support for PA management. We also acknowledge the role of pharmacotherapy (GLP-1 agonists and GIPs) in clinical care for patients with overweighr and obesity, and the added support these patients may need. The investigative team proposes a reimbursable service of a health coach to work collaboratively with PCPs, to deliver a Fitbit-supported PA program to patients with overweight/obesity who have been prescribed a weight loss medication. In Aim 1, the team will enroll PCPs to refer patients to a 12-week health coaching program. In Aim 2, the team will conduct interviews with enrolled patients/PCPs to understand their perspectives on the program, and with new sites to establish relationships for a future R01 submission.

DETAILED DESCRIPTION:
In Aim 1, after the patient has signed consent with the study coordinator, the coordinator will schedule the patient for their baseline in-person visit, and a flowsheet for the fitness tracker will be placed in the EHR by the study clinicians. During the baseline visit, the study team will assess height and weight, waist circumference assessment, and body composition. The 3-month follow-up visit will include the same measurements as listed above. Once baseline measures are completed, patients without a Fitbit device will be provided one for the duration of the study, which they get to keep. The same option will be available for patients who already have a Fitbit but would like one provided by the study team anyway. Patients will also install the Fitbit application and MyChart application (if needed) and sync the Fitbit with their patient portal with direction from the study team. Participants will also be instructed to wear their Fitbit for a total of 12 weeks. They will be provided a suggested step count to be accomplished from the health coach once they meet for the first session

Patients will have their first meeting scheduled with the health coach (up to 60-minutes in length, remotely). Patients will then meet with the health coach up to 5 more times (remotely) for up to 30-minutes per session over the course of the 12 weeks in the study. Health coaches will schedule meetings with the patients and communicate via Mychart. All sessions will be telehealth, conducted and recorded over Zoom. Patients will participate in the study for up to 12 weeks. Patients will receive support from the study team during the study period to troubleshoot any device related issue.

In Aim 2, patients and providers will provide verbal consent and be interviewed by the study research coordinator to assess workflow acceptability, perceptions, areas for workflow modification, preferences for initial training, preferences for frequency of review of remote monitoring data, and health coach interactions. The study team will interview patients during and at the completion of their 12 weeks to understand their perceptions on the program and supports needed, such as activity goals, feedback etc. Interviews will be 30-minutes in length, audio recorded only.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥27-45
* Prescribed a GLP-1/GIP within the past 6 months
* Currently taking GLP/GIP
* Age 18 years of age and older
* Patient of UMass Medical Group Primary Care Clinic
* Speaks and reads English

Exclusion Criteria:

* BMI <27 or ≥45
* Not currently taking GLP-1/GIP
* Under 18 years of age
* Prescribed GLP-1/GIP for less than 6 months
* Not a patient of UMass Medical Group Primary Care Clinic
* Does not speak English

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of enrollment | 6-months
  The number of enrolled patients in the study.

SECONDARY OUTCOMES:
Engagement with intervention | 3-months
  The proportion of scheduled visits the patient completes with the health coach over the 3-month study.
Average steps per day | Baseline, 3-months
  The average steps per day over the course of 1-week.
Short-Form 12 Question Health-related Quality of Life | Baseline, 3-months
  12-item self-report survey assessing quality of life. Scores range from 0-100 with a higher score indicating more positive health-related quality of life.
Numeric Pain Rating Scale (NPRS) | Baseline, 3-months
  6-questions regarding pain in body parts and doing activities of daily living using a Likert Scale from 0 to 10. Scores range from 0 (minimum) to 50 (maximum) with higher scores indicating greater levels of pain.
Muscle Strengthening Activities | Baseline, 3-months
  The Muscle-Strengthening Exercise Questionnaire (MSEQ) is a 4-item questionnaire assessing the weekly frequency, session duration and intensity, types of MSE (e.g., weight machines, bodyweight exercise) and muscle groups targeted. Scores range from 0 (minimum) to 7 (maximum), with higher scores indicating higher frequency of muscle strengthening activities.
Short-form Dietary Recall | Baseline, 3-months
  A short-form 15-item Food Frequency Questionnaire (FFQ) is a dietary assessment tool designed to estimate an individual's usual intake of specific food groups over a given period. The scores range from 15 (minimum) to 75 (maximum), with higher scores indicating consumption of a healthier diet.
Self-Report Physical Activity (IPAQ-SF) | Baseline, 3-months
  The Physical Activity Questionnaire - Short Form (PAQ-SF) is a brief, self-reported questionnaire designed to assess an individual's physical activity levels over a specified period, typically the past 7 days. It is a condensed version of longer physical activity questionnaires, making it practical for use in research, clinical settings, and population health surveys. The minimum score is 0 (no minutes per week), and there is no maximum. Higher scores indicate higher levels of physical activity.
Exercise Self Efficacy | Baseline, 3-months
  A 24-item tool assessing barriers that get in the way of physical activity on a Likert scale of 1 to 5. The scores range from 24 (minimum) to 168 (maximum) with a higher score indicating greater exercise self-efficacy.
Eating Self-Efficacy Brief Scale | Baseline, 3-months
  Designed to assess an individual's confidence in their ability to control eating behaviors across different situations. It is rooted in self-efficacy theory, which emphasizes the role of belief in one's capability to perform specific behaviors. Consists of 7 items using a Likert scale of 1 to 5 for responses. The total score range is 10 (minimum) to 70 (maximum), with a higher score indicating greater eating self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year afte the study ends.
Access Criteria: We will share de-identified data upon reasonable request.